CLINICAL TRIAL: NCT03637725
Title: Multi-center Trial of SPECT Myocardial Blood Flow Quantitation for Detection of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: SPECT MBFQ Trial I
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease: Suspected or known coronary artery disease

SUMMARY:
Patients with suspected or known coronary artery disease who are scheduled for clinically indicated SPECT myocardial perfusion imaging (MPI) and will receive invasive coronary angiogram are recruited to receive SPECT MBF study.

DETAILED DESCRIPTION:
Patients with suspected or known coronary artery disease who are scheduled for clinically indicated SPECT myocardial perfusion imaging (MPI) and likely will further receive invasive coronary angiogram will be recruited for a SPECT MBF study. The MBF study will be performed as an adjunct to MPI utilizing the same rest and stress injections of 99mTc-Sestamibi (MIBI) tracer, and the same infusion of dipyridamole, adenosine or adenosine triphosphate for stressing. The MBF study will be completed in single or two days depending on the imaging protocol of MPI for a site. This is an observational study with no interventions to the clinical routine whatsoever. Three models of SPECT (GE NM530c) and SPECT/CT (Siemens Symbia-T16 and -T2) cameras are included to acquire rest/stress dynamic SPECT and MPI data. A CT scan will be acquired for the purpose of attenuation correction. All dynamic images will be reconstructed with physical corrections, including attenuation, scatter, resolution recovery and noise reduction, and processed to quantify MBF with the same kinetic modeling. The imaging processing of MBF study will be conducted with a SPECT MBF dedicated software (MyoFlowQ) in a central lab. MPI images will be collected and independently read by three consensus readers. The angiographic result will be independently reviewed by an interventional cardiologist. Diagnostic performance of SPECT MBF and perfusion will be compared utilizing angiographic result as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 79 years old
* Any CAD risk factor
* CAD related symptoms
* Intermediate to high probability of CAD
* Suspected or known CAD on a stable medication regime
* Able and willing to comply with the study procedures
* Written informed consent

Exclusion Criteria:

* History or risk of severe bradycardia
* History of myocardial infarction, dilated cardiomyopathy, hypertrophic cardiomyopathy, valve issue or congenital heart disease
* Wheezing asthma or COPD
* Known second- or third-degree AV block
* Known hypersensitivity to dipyridamole or adenosine
* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult male and female patients who have suspected or known CAD are agreed to receive MBF measurements when their MPI scan will be performed clinically.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of MBF and MPI | Through the study completion up to 12 months
  The diagnostic accuracy of MBF and MPI while angiography is utilized as the reference standard

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, MD/PhD, Study Chair — Fu Wai Hospital, Beijing, Chia; Jianming Li, MD/PhD, Principal Investigator — TEDA International Cardiovascular Hospital; Yuming Zheng, MD, Principal Investigator — China-Japanese Friendship Hospital, Beijing, China; Jie Zhang, MD/MS, Principal Investigator — Central China Fuwai Hospital, Henan, China
Locations (4):
- China (4):
  - China-Japanese Friendship Hospital, Beijing
  - Fuwai Hospital, Beijing
  - Teda International Cardiovascular Hospital, Tanjin
  - Central China Fuwai Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang L, Zheng Y, Zhang J, Wang M, Wu D, Wang Y, Qiu H, Hsu B, Fang W. Diagnostic value of quantitative myocardial blood flow assessment by NaI(Tl) SPECT in detecting significant stenosis: a prospective, multi-center study. J Nucl Cardiol. 2023 Apr;30(2):769-780. doi: 10.1007/s12350-022-03085-3. Epub 2022 Aug 15. PMID 35971031